CLINICAL TRIAL: NCT00106288
Title: A Multicenter, Double Blind, Comparative, Randomized Study to Evaluate the Efficacy and Safety of Micafungin (FK463) Versus Liposomal Amphotericin B (AmBisome) in the Treatment of Invasive Candidiasis and Candidemia
Brief Title: Micafungin Versus AmBisome in Invasive Candidiasis and Candidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FG-463-21-08
Record Dates: First submitted 2005-03-22; First posted 2005-03-23 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Candidiasis
Keywords: Candidaemia; Micafungin
MeSH Terms: conditions — Candidiasis; Candidemia | interventions — Micafungin; liposomal amphotericin B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Micafungin
- 2 (Active Comparator)
  Interventions: Drug: Liposomal Amphotericin B

INTERVENTIONS:
Drug: Micafungin — IV
  Other Names: Mycamine; FK463
  Arms: 1
Drug: Liposomal Amphotericin B — IV
  Other Names: AmBisome
  Arms: 2

SUMMARY:
The purpose of this study is to determine the efficacy and safety of micafungin (FK463) versus liposomal amphotericin B (AmBisome) in treating neutropenic and non-neutropenic patients with confirmed invasive candidiasis or candidemia. Enrollment will include adult and pediatric patients.

DETAILED DESCRIPTION:
A phase III, multicenter, double-blind, comparative, parallel, randomized study. Enrollment will include adult and pediatric patients. The adult population is sized to test for non-inferiority. For the pediatric population, descriptive analyses are planned.

ELIGIBILITY:
Inclusion Criteria:

Patients either non-neutropenic with absolute neutrophil counts >= 500 cells/mm3 or neutropenic with absolute neutrophil counts < 500 cells/mm3 must have:

* Candidemia or invasive candidiasis,
* Confirmation and typical clinical signs and symptoms by fungal culture and/or histology,
* Positive culture obtained no more than four days prior to the first dose of study medication.

Exclusion Criteria:

* Patient is pregnant or nursing
* Patients with evidence of liver disease as defined by: a) SGOT/AST or SGPT/ALT > 10 times the upper limit of normal (ULN); or b) Total bilirubin > 5 times ULN.
* Patients whose sole diagnosis is oropharyngeal and/or esophageal candidiasis and/or with positive cultures of urine specimens, sputum specimens, bronchoalveolar-lavage specimens or samples from indwelling drains.
* Patients who have received prophylactic/empiric therapy with azoles or conventional amphotericin B for more than three days within one week prior to enrollment. Neutropenic patients, however, may have received prophylactic azoles without time restrictions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2003-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Investigator's assessment of overall treatment success. Success is defined as clinical (complete or partial) and mycological (eradication or presumed eradication) response at the End of Therapy. | 6 and 12 weeks post treatment

SECONDARY OUTCOMES:
Clinical response (complete, partial, stabilization, progression) during the treatment period and the post-treatment period | During the 2 to 8 week treatment period and the 12 week post treatment followup period
Mycological response (eradication, presumed eradication, persistence) during the treatment period and the post-treatment period | During the 2 to 8 week treatment period and the 12 week post treatment followup period
Overall incidence of emergent and recurrent fungal infections at the End of Study | End of the 12 week post treatment followup peroid
Independent Efficacy Review Committee's assessment of overall treatment success | Prior to database lock
Peak change of estimated glomerular filtration rate during the treatment period compared to Baseline | During the 2 to 8 week treatment period
Incidence of acute infusion related reactions as pre-defined | During the 2 to 8 week treatment period
Patient survival at the End of Therapy and at the End of Study | End of the 2 to 8 week treatment period and end of the 12 week post treatment followup period
Overall incidence of Adverse Events (AE) | Throughout study and post treatment followup period

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (31):
- United States (22):
  - Birmingham, Alabama
  - Orange, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Hinsdale, Illinois
  - Maywood, Illinois
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - New York, New York
  - Rochester, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - San Antonio, Texas
  - Provo, Utah
- Canada (9):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Regina, Saskatchewan

REFERENCES:
- [Background] Kuse ER, Chetchotisakd P, da Cunha CA, Ruhnke M, Barrios C, Raghunadharao D, Sekhon JS, Freire A, Ramasubramanian V, Demeyer I, Nucci M, Leelarasamee A, Jacobs F, Decruyenaere J, Pittet D, Ullmann AJ, Ostrosky-Zeichner L, Lortholary O, Koblinger S, Diekmann-Berndt H, Cornely OA; Micafungin Invasive Candidiasis Working Group. Micafungin versus liposomal amphotericin B for candidaemia and invasive candidosis: a phase III randomised double-blind trial. Lancet. 2007 May 5;369(9572):1519-1527. doi: 10.1016/S0140-6736(07)60605-9. PMID 17482982
- [Background] Queiroz-Telles F, Berezin E, Leverger G, Freire A, van der Vyver A, Chotpitayasunondh T, Konja J, Diekmann-Berndt H, Koblinger S, Groll AH, Arrieta A; Micafungin Invasive Candidiasis Study Group. Micafungin versus liposomal amphotericin B for pediatric patients with invasive candidiasis: substudy of a randomized double-blind trial. Pediatr Infect Dis J. 2008 Sep;27(9):820-6. doi: 10.1097/INF.0b013e31817275e6. PMID 18679151
- [Background] Horn DL, Ostrosky-Zeichner L, Morris MI, Ullmann AJ, Wu C, Buell DN, Kovanda LL, Cornely OA. Factors related to survival and treatment success in invasive candidiasis or candidemia: a pooled analysis of two large, prospective, micafungin trials. Eur J Clin Microbiol Infect Dis. 2010 Feb;29(2):223-9. doi: 10.1007/s10096-009-0843-0. Epub 2009 Dec 15. PMID 20013016
- [Derived] Shorr AF, Wu C, Kothari S. Outcomes with micafungin in patients with candidaemia or invasive candidiasis due to Candida glabrata and Candida krusei. J Antimicrob Chemother. 2011 Feb;66(2):375-80. doi: 10.1093/jac/dkq446. Epub 2010 Dec 8. PMID 21147825
- [Derived] Dupont BF, Lortholary O, Ostrosky-Zeichner L, Stucker F, Yeldandi V. Treatment of candidemia and invasive candidiasis in the intensive care unit: post hoc analysis of a randomized, controlled trial comparing micafungin and liposomal amphotericin B. Crit Care. 2009;13(5):R159. doi: 10.1186/cc8117. Epub 2009 Oct 5. PMID 19804626